CLINICAL TRIAL: NCT05717933
Title: Thyroid Function Among Pediatric Patients With Type 1 Diabetes Mellitus at Firs Presentation, From Patients' Characteristics to Disease Severity
Brief Title: Thyroid Function Among Pediatric Patients With DM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Fathy Abd ELhay, Principal Investigator, Assiut University
Other Study IDs: thyroid function in DM
Record Dates: First submitted 2022-09-01; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Thyroid Function in DM

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: thyroid hormones — Thyroid function among pediatric patients with type1 diabetes mellitus at the first presentation, from patients' characteristics to disease severity

SUMMARY:
Thyroid function among pediatric patients with type1 diabetes mellitus at the first presentation, from patients' characteristics to disease severity

DETAILED DESCRIPTION:
Type-I diabetes mellitus is an auto immune disease. It is the most common type of diabetes in children and adolescents. It is also the most common chronic disease in children in the developed countries. The illness is characterized by the body's inability to produce insulin due to the autoimmune destruction of the beta cells in the pancreas. Globally, it is estimated that there are almost 500,000 children aged under 15 years with type 1diabetes, with large geographical variations in incidence.

* Furthermore Between 10 to 70% of these children present in Diabetic Ketoacidosis (DKA) as their first presentation of the disease.
* In addition It can be associated with other auto immune disorders that may influence the control of diabetes by disruption of the function of respective organs and enhance the opportunity of developing DKA as the first manifestation of their disease.
* In particular, autoimmune thyroiditis (AIT) is the most common disorder associated with type 1 Diabetes Mellitus.
* AIT and type 1 Diabetes Mellitus have a common genetic background and similar pathogenesis; hence, they could occur in the same individual or family. The prevalence of thyroid autoantibodies in children with type1 Diabetes Mellitus ranges from 3% to 50% in different countries and populations, which is markedly higher than in the general population (range, 1% to 4%).
* Besides thyroid autoantibodies can be detected at the initial diagnosis and after it.
* Thyroiditis is often clinically silent but it may progress to autoimmune thyroid disease (AITD), recognized as overt or subclinical hypothyroidism or hyperthyroidism.
* The American Diabetes Association (ADA) recommended screening Thyroid-Stimulating hormone after diagnosis of diabetes and then after every one to two years. It also recommended that patients found to have positive anti-Thyroid Peroxidase antibodies with normal thyroid function tests should be screened more frequently, every six months to a year .

ELIGIBILITY:
Inclusion Criteria:

* - patients between 2 year and <18 years of age in both sex
* patients with T1DM that had not been on any thyroid medication

Exclusion Criteria:

* - patients <2 years and >18 years of age in both sex
* patient with systemic illnesses, diagnosed thyroid disorders and patients taking medications

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Type-I diabetes mellitus is an auto immune disease. It is the most common type of diabetes in children and adolescents. It is also the most common chronic disease in children in the developed countries. The illness is characterized by the body's inability to produce insulin due to the autoimmune destruction of the beta cells in the pancreas. Globally, it is estimated that there are almost 500,000 children aged under 15 years with type 1diabetes, with large geographical variations in incidence[1].
  * Furthermore Between 10 to 70% of these children present in Diabetic Ketoacidosis (DKA) as their first presentation of the disease[2].
  * In addition It can be associated with other auto immune disorders that may influence the control of diabetes by disruption of the function of respective organs and enhance the apportunity of developing DKA as the first manifestation of their disease. [3,4]
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
thyroid abnormalities among children and adolescents with type 1 diabetes mellitus when its first detected and its relationship with disease-related variables. | Baseline
  The aim of this study was to detect the prevalence of thyroid functions TSH,T3,T4 abnormalities and the relationship of positive anti-thyroid antibodies to potential risk factors, including, age, gender, duration of diabetes among children and adolescents with type 1 diabetes mellitus when its first detected

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Metwalley KA, El-Saied AR. Thyroid abnormalities in Egyptian children and adolescents with type 1 diabetes mellitus: A single center study from Upper Egypt. Indian J Endocrinol Metab. 2014 Sep;18(5):637-41. doi: 10.4103/2230-8210.139218. PMID 25285279